CLINICAL TRIAL: NCT02903251
Title: Acute and Long-term Effects of Intranasal Oxytocin in Alcohol Withdrawal and Dependence: A Prospective Randomized Parallel Group Placebo-controlled Trial
Brief Title: Oxytocin and Alcohol Withdrawal and Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Lade Addiction Treatment Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 140682; 2015-004463-37 (EudraCT Number)
Record Dates: First submitted 2016-08-30; First posted 2016-09-16 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Alcoholism; Substance-Related Disorders
Keywords: Oxytocin; Administration, Intranasal; Ethanol
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin (Experimental): intranasal oxytocin spray Day 1-3: Twice daily intranasal oxytocin spray administered by health personnel.
  Day 3-30: Self-administered intranasal spray as needed, max thrice daily intranasal spray without oxytocin
  Interventions: Drug: intranasal oxytocin spray
- Placebo (Placebo Comparator): intranasal spray without oxytocin Day 1-3: Twice daily intranasal spray without oxytocin, administered by health personnel.
  Day 3-30: Self-administered intranasal spray as needed, max thrice daily
  Interventions: Other: intranasal spray without oxytocin

INTERVENTIONS:
Drug: intranasal oxytocin spray — 6 insufflations (24 IU of oxytocin total) given twice daily, day 1-3. 2 insufflations (8 IU of oxytocin total) as needed, max thrice daily, day 3-30.
  Other Names: Syntocinon
  Arms: oxytocin
Other: intranasal spray without oxytocin — 6 insufflations (24 IU of placebo total) given twice daily, day 1-3. 2 insufflations (8 IU of placebo total) as needed, max thrice daily, day 3-30.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This study evaluates the effect of oxytocin nasal spray on alcohol withdrawal and dependence in adults admitted for detoxification of alcohol, and during the following 4 weeks in an outpatient setting. Half of the participants will receive oxytocin nasal spray, the other half placebo nasal spray.

ELIGIBILITY:
Inclusion Criteria:

1. At least one prior episode 2 days or longer in duration during which the subject experienced withdrawal symptoms that caused significant incapacitation (e.g., inability to work or do normal activities) OR at least one prior inpatient or outpatient medical detoxification during which the subject exhibited withdrawal symptoms of sufficient magnitude that sedative-hypnotic or anticonvulsant medication was required at least once on 2 consecutive days after cessation of or reduction in the use of alcohol following 2 weeks or more of heavy daily consumption
2. average consumption of 8-30 standard drinks per day for at least 2 weeks prior to enrollment in the study;
3. consenting to participate in the study;
4. have residency in Trøndelag County after discharge

Exclusion Criteria:

1. chronic treatment with sedative-hypnotic medications such as benzodiazepines or z-hypnotics;
2. dependence on substances other than alcohol, nicotine or caffeine;
3. inadequately treated, unstable and/or compromising medical or psychiatric conditions;
4. low body weight (BMI < 17) or history of anorexia nervosa or bulimia in the past 2 years;
5. pregnancy; parturition or breast-feeding in the past 6 months;
6. inability to read well enough to complete study questionnaires determined by whether the prospective subject can read the consent form without help and correctly answer basic questions about information in the consent form;
7. no alcohol in the blood and > 15 h since last intake of alcohol;
8. prior inclusion and participation in the same study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Total oxazepam dosage in milligrams | 3 days
  total oxazepam dosage per subject during detoxification, as determined by Clinical Institute Withdrawal Assessment-Alcohol, Revised (CIWA-Ar) scores
Alcohol intake | 30 days
  Alcohol intake of outpatients, using blood, urine, Timeline Followback and diaries.

SECONDARY OUTCOMES:
Sleep | 3 days
  self-reported sleeping hours
Sleep | 30 days
  self-reported sleeping hours
motor activity | 3 days
  assessed by actigraph
alcohol craving | day 3
  self-reported using Alcohol Craving questionnaire short form revised, Norwegian version (ACQ-SF-R)
alcohol craving | day 30
  self-reported using Alcohol Craving questionnaire short form revised, Norwegian version (ACQ-SF-R)
Mental distress | day 3
  measured by Hopkins Symptoms Checklist 10 items (SCL-10)
Mental distress | day 30
  measured by Hopkins Symptoms Checklist 10 items (SCL-10)
patient activity | day 3
  measured by Patient Activity Measure 13 (PAM-13)
patient activity | day 30
  measured by Patient Activity Measure 13 (PAM-13)
Socio-emotional recognition | Day 2
  assessed by Reading the mind in the eyes test (RMET)
Socio-emotional recognition | Day 3
  assessed by Reading the mind in the eyes test (RMET)
Socio-emotional recognition | day 30
  assessed by Reading the mind in the eyes test (RMET)
Facial emotional selective attention | Day 2
  assessed by Visual Dot probe task
Facial emotional selective attention | Day 3
  assessed by Visual Dot probe task
Facial emotional selective attention | day 30
  assessed by Visual Dot probe task

CONTACTS AND LOCATIONS:
Overall Officials: Trond Jacobsen, MD PhD, Study Director — St Olav's University Hospital Trondheim; Olav Spigset, MD PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Lade Addiction Treatment Center, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Melby K, Grawe RW, Aamo TO, Salvesen O, Spigset O. Effect of intranasal oxytocin on alcohol withdrawal syndrome: A randomized placebo-controlled double-blind clinical trial. Drug Alcohol Depend. 2019 Apr 1;197:95-101. doi: 10.1016/j.drugalcdep.2019.01.003. Epub 2019 Feb 13. PMID 30784955